CLINICAL TRIAL: NCT02353858
Title: Preoperative Radiochemotherapy With Concurrent Deep Regional Hyperthermia for Locally Advanced Rectal Cancer. A Prospective Phase II Trial
Brief Title: Preoperative Radiochemotherapy With Hyperthermia for Locally Advanced Rectal Cancer
Acronym: HT01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HT01
Record Dates: First submitted 2014-12-02; First posted 2015-02-03 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Rectal Cancer; Locally Advanced Rectal Cancer; Hyperthermia; Hyperthermic Radiochemotherapy; Hyperthermic Chemoradiotherapy; Deep Regional Hyperthermia
Keywords: Rectal Cancer; Hyperthermia; Radiochemotherapy; Chemoradiotherapy; Deep regional hyperthermia; pathologic complete response; Regression Grade; Locally advanced rectal cancer; complete response
MeSH Terms: conditions — Rectal Neoplasms; Hyperthermia; Pathologic Complete Response | interventions — Radiotherapy; Drug Therapy; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RtChx + Hyperthermia (Experimental): Radiotherapy: 5 x 1,8 Gy/Week, cumulative dose 50,4 Gy (ICRU) Chemotherapy: 5-fluorouracil d1-5 and d29-d33 Deep regional hyperthermia: 2x/week
  Interventions: Other: Deep regional hyperthermia; Radiation: Radiotherapy; Drug: Chemotherapy (5-Fluorouracil)

INTERVENTIONS:
Other: Deep regional hyperthermia — Deep regional hyperthermia of the pelvis, Total time 90 min, Target temperature 41-42°C.
Radiation: Radiotherapy — Radiotherapy of the primary tumor and pelvis, 5 x 1,8 Gy per week, total Dose: 50,4 Gy.
Drug: Chemotherapy (5-Fluorouracil) — 5-Fluorouracil, continuous venous infusion week 1 and 5. 1000 mg per square meter of body-surface area per day.

SUMMARY:
The current trial is evaluating the impact of deep regional hyperthermia on the pathological complete response rate in locally advanced rectal cancer in the context of preoperative 5FU based radiochemotherapy.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed Adenocarcinoma of the rectum (up to 10 cm from the anal verge)
* International Union Against Cancer stages II or III
* ECOG PS 0/2
* Informed consent

Exclusion Criteria:

* Congestive heart failure (NYHA III/IV)
* History of myocardial infarction within the last 6 months.
* AV Block III
* Total hip replacement or major metal pelvic implants
* Cardiac pacemaker
* Contraindications for radiochemotherapy
* Contraindications for surgical tumor resection
* Previous pelvic radiotherapy or chemotherapy
* Active chronic inflammatory bowel disease
* Collagenosis
* Congenital diseases with increased radiosensitivity
* Pregnancy or breastfeeding
* Secondary malignancies other than locally controlled basalioma or in-situ carcinomas Infiltration of the anal canal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-08; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Pathological complete response rate | After surgical resection (4-6 weeks after last radiotherapy fraction)

SECONDARY OUTCOMES:
Locoregional progression free survival | 3 years
Disease free survival | 3 years
Distant metastases free survival | 3 years
Overall survival | 3 years
Number of hyperthermia treatments | At completion of hyperthermic radiochemotherapy
Acute and chronic treatment related toxicity, according to CTC criteria | 3 years
post operative morbidity | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tübingen, Department of Radiation Oncology, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Gani C, Lamprecht U, Ziegler A, Moll M, Gellermann J, Heinrich V, Wenz S, Fend F, Konigsrainer A, Bitzer M, Zips D. Deep regional hyperthermia with preoperative radiochemotherapy in locally advanced rectal cancer, a prospective phase II trial. Radiother Oncol. 2021 Jun;159:155-160. doi: 10.1016/j.radonc.2021.03.011. Epub 2021 Mar 17. PMID 33741467